CLINICAL TRIAL: NCT05207384
Title: Comparison of Ultrasound-Guided Subacromial Ozone (O2-O3) and Corticosteroid Injections in the Treatment of Chronic Rotator Cuff Tendinopathy: A Randomized Controlled Trial
Brief Title: Comparison of Subacromial Ozone (O2-O3) and Corticosteroid Injections in the Treatment of Rotator Cuff Tendinopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gaziler Physical Medicine and Rehabilitation Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Yasin Demir, Physical Medicine and Rehabilitation Associate Professor, Gaziler Physical Medicine and Rehabilitation Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 26
Record Dates: First submitted 2021-12-25; First posted 2022-01-26 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-06

CONDITIONS: Rotator Cuff Tendinopathy
Keywords: rotator cuff tendinopathy; ozone; steroid; ultrasonography
MeSH Terms: interventions — Ozone; Injections; Adrenal Cortex Hormones

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcome measures will be evaluated by an independent physiatrist, blinded for the assigned treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ozone (O2-O3) group (Active Comparator): Ultrasound (US)-guided injections will be performed with a 5-12 MHz linear transducer (Logic e portable; GE Healthcare, China) by the same physiatrist and injections will be administered into the subacromial bursa with a posterolateral approach. 3 sessions (1 session/week) of 5 mL of ozone (O2-O3) will be injected (with a concentration of 10 μg/mL in the first session, 15 μg/mL in the second session, and 20 μg/mL in the third session).
  Interventions: Procedure: Ozone (O2-O3) injection
- Corticosteroid group (Other): US-guided injection will be performed with a 5-12 MHz linear transducer (Logic e portable; GE Healthcare, China) by the same physiatrist and injections will be administered into the subacromial bursa with a posterolateral approach. A mixture of 1 mL corticosteroid (betamethasone 3 mg/mL) and 1 mL lidocaine (20 mg) will be injected (1 session).
  Interventions: Procedure: Corticosteroid injection

INTERVENTIONS:
Procedure: Ozone (O2-O3) injection — US-guided injections will be performed with a 5-12 MHz linear transducer (Logic e portable; GE Healthcare, China) by the same physiatrist and injections will be administered into the subacromial bursa with a posterolateral approach. 3 sessions (1 session/week) of 5 mL of ozone (O2-O3) will be injected (with a concentration of 10 μg/mL in the first session, 15 μg/mL in the second session, and 20 μg/mL in the third session).
  Arms: Ozone (O2-O3) group
Procedure: Corticosteroid injection — US-guided injections will be performed with a 5-12 MHz linear transducer (Logic e portable; GE Healthcare, China) by the same physiatrist and injections will be administered into the subacromial bursa with a posterolateral approach. A mixture of 1 mL corticosteroid (betamethasone 3 mg/mL) and 1 mL lidocaine (20 mg) will be injected (1 session).
  Arms: Corticosteroid group

SUMMARY:
Shoulder pain accounts for approximately 16% of all musculoskeletal symptoms. Rotator cuff tendinopathy is the most common cause of shoulder pain.

The aim of this study is to compare the effects of ultrasound-guided subacromial ozone (O2-O3) versus corticosteroid injection in patients with chronic rotator cuff tendinopathy.

DETAILED DESCRIPTION:
Shoulder pain accounts for approximately 16% of all musculoskeletal symptoms. Rotator cuff tendinopathy is the most common cause of shoulder pain.

There are limited studies comparing the efficacy of ozone and corticosteroid injections in rotator cuff tendinopathy. In this context, the aim of this study is to compare the effects of ultrasound-guided subacromial ozone (O2-O3) versus corticosteroid injection in patients with chronic rotator cuff tendinopathy.

ELIGIBILITY:
Inclusion Criteria:

* aged between 18 and 70 years
* pain in the shoulder region and increase in pain with overhead-throwing activity
* chronic shoulder pain for more than 3 months
* partial rotator cuff tear or rotator cuff tendinosis diagnosed by US or magnetic resonance imaging (MRI).

Exclusion Criteria:

* a full-thickness rotator cuff tear diagnosed by US or MRI
* allergic reaction betamethasone or lidocaine
* contraindications for ozone (O2-O3) injection, such as uncontrolled hyperthyroidism, glucose-6 phosphate dehydrogenase deficiency (G6PDD), pregnancy and platelet level <50 103/µL
* history of coagulopathy, diabetes, or hepatitis
* intra-articular/subacromial injections in the last 3 months
* history of shoulder infection, fracture, trauma, bony lesion, tumor or inflammatory rheumatic diseases
* history of brachial plexus lesion/cervical radiculopathy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2022-01-27 (Actual); Primary Completion 2022-05-20 (Actual); Study Completion 2022-05-20 (Actual)

PRIMARY OUTCOMES:
The Western Ontario Rotator Cuff Index (WORC) | at baseline and change from baseline WORC at 4 weeks and 12 weeks after injections
  The Western Ontario Rotator Cuff Index (WORC) is a self-administered assessment tool for rotator cuff disease. WORC has 21 questions in 5 domains consisting of work, physical symptoms, social well-being, emotional well-being, and sports and recreation. Each question is scored on a 100-mm, with higher scores demonstrating larger problems. Turkish validity of the WORC has been illustrated.

SECONDARY OUTCOMES:
The Shoulder Pain and Disability Index (SPADI) | at baseline and change from baseline SPADI at 4 weeks and 12 weeks after injections
  The Shoulder Pain and Disability Index (SPADI) is a 13 item self-assessment measurement tool to evaluate disability (8 items) and pain (5 items). The subscales of disability and pain are measured as the average of the corresponding items between 0-100, with higher scores indicating greater disability and pain.
Visual Analogue Scale (VAS) | at baseline and change from baseline VAS at 4 weeks and 12 weeks after injections
  The severity of the patients' shoulder pain in the last week will be evaluated using the 10-point VAS (from 0 (no pain) to 10 (worst imaginable pain))

OTHER OUTCOMES:
Ultrasonographic measurements | at baseline and change from baseline ultrasonographic measurements at 4 weeks and 12 weeks after injections
  supraspinatus tendon thickness, subacromial bursa thickness and acromiohumeral distance will be measured by US in both groups

CONTACTS AND LOCATIONS:
Locations (1):
- Merve Örücü Atar, Ankara, Cankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No